CLINICAL TRIAL: NCT03319888
Title: Effect of CPAP in the Worsening of Renal Function in Early Stages of Chronic Kidney Disease (CKD)
Acronym: Renas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Jaime Corral Penafiel, Principal Investigator, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI15/00137
Record Dates: First submitted 2016-09-23; First posted 2017-10-24 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2017-10

CONDITIONS: Chronic Kidney Insufficiency; Sleep Apnea
Keywords: CPAP, Chronic kidney disease, sleep apnea
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sleep Apnea Syndromes; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Conservative Treatment

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cpap group (Experimental): CPAP treatment plus conservative treatment with lifestyle modifications.
  Interventions: Device: CPAP
- control group (Active Comparator): Conservative treatment with lifestyle modifications.
  Interventions: Other: conservative treatment

INTERVENTIONS:
Device: CPAP — continuous positive pressure in the airway
  Arms: cpap group
Other: conservative treatment — conservative treatment group with lifestyle modifications
  Arms: control group

SUMMARY:
Objectives: Evaluate the effect of CPAP to reduce the progression of chronic kidney disease or CKD (the decline of glomerular filtration rate is ≥ 30%) in patients with early-stage renal disease and sleep apnea syndrome (OSAS). Other objectives are; determine the prevalence of OSAS in patients with early-stage renal disease and evaluate the changes in inflamatories markers and endothelial damage, the state of KDIGO, cardiovascular events, mortality and cost-effectiveness analysis in CPAP group versus non-CPAP group patients.

Methods: A prospective, multicentric, randomized and controlled study will be carried out for 3 years. Early-stage renal disease (G1-3 KDIGO) and OSAS patients will be included. The investigators will make a respiratory polygraphy to determinate OSAS (AHI ≥15/h) and after that, the investigators randomized patients in 2 groups; CPAP group and control group (non-CPAP treatment). Patients with AHI <15/h (non-OSAS) will be the reference group and the half of these patients, randomly chosen, will be followed up at the end of the follow up.

Statistic analysis: the investigators will analyze the differences in glomerular filtration rate before and after the treatment, comparing the percentage of patients with CKD progression for both groups. The investigators will use the chi square test with raw data and adjusted for confounding variables using intention to treat analysis with imputation of missing values.

DETAILED DESCRIPTION:
There is a bidirectional involvement between the chronic kidney disease (CKD) and sleep apnea syndrome (OSAS). The declining of renal function, the fluid overloading and the disturbance of ventilation control could cause sleep apneas. On the other hand, the nocturnal hypoxia in patients with OSAS has been associated with changes in the renin-angiotensin system and sympathetic nervous system and production of reactive oxygen species. These findings are relationed with the deterioration of kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the outpatient nephrology department with a diagnosis of chronic kidney disease stages G1-3 KDIGO
* Older than18 years
* Habitual snoring or observed apneas
* Scale sleep sleepiness (Epworth Test) with 11 points or lower.

Exclusion Criteria:

* Very debilitating chronic or neoplastic disease
* Respiratory failure (PaO 2 <55 mm Hg).
* Other symptoms of suspected sleep disorder different from OSAS.
* Patients unable to perform self-administered questionnaires.
* Patients with> 50% of central apnea or Cheyne-Stokes.
* Patients who do not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-11-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
To test whether treatment with CPAP in patients with moderate to severe OSAS and CKD in stages KDIGO G1-3, reduces the progression of renal disease (30% drop in GF) after 2 years of followed up. | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  Number of participants with chronic kidney disease (CKD) and obstructive sleep apnea syndrome (OSAS) with a 30% decline in estimated glomerular filtration rate (eGFR) using the CKD-EPI (CKD Epidemiology Collaboration) 2009 creatinine equation after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)

SECONDARY OUTCOMES:
To estimate the prevalence of OSAS in patients with CKD stages G1-3 KDIGO | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  Number of participants with CKD and snoring and observed apneas with an apnea and hypoapnea index (AHI) ≥15/hour in home-based polysomnography.
To test whether treatment with CPAP reduces the albumin / creatinine ratio in urine. | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  Number of participants with CKD and OSAS with a decline in urine albumin to creatinine ratio.
To evaluate whether treatment with CPAP reduces serum Cystatin C | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  Number of participants with CKD and OSAS with a decline in serum cystatin C levels
To evaluate whether treatment with CPAP reduces inflammation-endothelial disfunction markers | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  Number of participants with CKD and OSAS with a decline in inflammation-endothelial disfunction markers (interleukine-6, interleukine-8, reactive C protein, sedimentation rate, asymmetric dimethylaginine or ADMA, intercellular adhesion molecule 1 or ICAM-1, vascular adhesion protein 1 or VCAM 1, vascular endothelial growth factor or VEGF)
Evaluate whether treatment with CPAP reduces the progression of CKD to a different stage | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  number of participants with CKD and OSAS with a change to a higher CKD stage according to eGFR.
to test wheather CPAP reduces the percentage of patients achieving replacement therapy | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  number of participants with CKD and OSAS who need renal replacement therapy (haemodialysis, peritoneal dialysis or renal transplantation)
Evaluate wheather treatment with CPAP reduces the incidence of cardiovascular events | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  number of participants with CKD and OSAS who suffered a cardiovascular event (myocardial infarction, stroke, hospitalization for heart failure, atrial fibrillation)
Evaluate wheather treatment with CPAP reduces the mortality | after 2 years of followed up (each patient will be followed up for at least 2 years - range from 2 to 3 years)
  number of participants with CKD and OSAS with CPAP treatment who died (all-cause mortality)
Evaluation of the cost-effectiveness of treatment groups with and without CPAP | after 2 years of followed up (each patient will be followed up for at least 2 years-range from 2 to 3 years)
  Cost-effectiveness of treatment groups conducting a cost-effectiveness study that allow us to estimate the incremental cost-effectiveness ratio (ICER) of CPAP treatment group compared to the conventional treatment group
Compare the evolution of inflammation-endothelial disfunction markers in NO-OSAS group versus OSAS group | after 2 years of followed up (each patient will be followed up for at least 2 years-range from 2 to 3 years)
  Number of participants with NO-OSAS versus OSAS who have a decline in inflammation-endothelial disfunction markers (interleukine-6, interleukine-8, reactive C protein, sedimentation rate, asymmetric dimethylaginine or ADMA, intercellular adhesion molecule 1 or ICAM-1, vascular adhesion protein 1 or VCAM 1, vascular endothelial growth factor or VEGF)
Compare the worsening of the glomerular filtration in NO OSAS group versus OSAS group | after 2 years of followed up (each patient will be followed up for at least 2 years-range from 2 to 3 years)
  number of participants with NO OSAS versus OSAS who have a worsening of the glomerular filtration.
Compare the percentage of patients achieving renal replacement therapy in NO OSAS group versus OSAS group | after 2 years of followed up (each patient will be followed up for at least 2 years-range from 2 to 3 years)
  number of participants who need renal replacement therapy in NO OSAS group versus OSAS group

CONTACTS AND LOCATIONS:
Locations (1):
- Jaime Corral, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha V, Garcia-Garcia G, Iseki K, Li Z, Naicker S, Plattner B, Saran R, Wang AY, Yang CW. Chronic kidney disease: global dimension and perspectives. Lancet. 2013 Jul 20;382(9888):260-72. doi: 10.1016/S0140-6736(13)60687-X. Epub 2013 May 31. PMID 23727169
- [Background] James MT, Hemmelgarn BR, Tonelli M. Early recognition and prevention of chronic kidney disease. Lancet. 2010 Apr 10;375(9722):1296-309. doi: 10.1016/S0140-6736(09)62004-3. PMID 20382326
- [Background] Otero A, de Francisco A, Gayoso P, Garcia F; EPIRCE Study Group. Prevalence of chronic renal disease in Spain: results of the EPIRCE study. Nefrologia. 2010;30(1):78-86. doi: 10.3265/Nefrologia.pre2009.Dic.5732. Epub 2009 Dec 14. PMID 20038967
- [Background] Lloberes P, Duran-Cantolla J, Martinez-Garcia MA, Marin JM, Ferrer A, Corral J, Masa JF, Parra O, Alonso-Alvarez ML, Teran-Santos J. Diagnosis and treatment of sleep apnea-hypopnea syndrome. Spanish Society of Pulmonology and Thoracic Surgery. Arch Bronconeumol. 2011 Mar;47(3):143-56. doi: 10.1016/j.arbres.2011.01.001. No abstract available. English, Spanish. PMID 21398016
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Nicholl DDM, Ahmed SB, Loewen AHS, Hemmelgarn BR, Sola DY, Beecroft JM, Turin TC, Hanly PJ. Declining kidney function increases the prevalence of sleep apnea and nocturnal hypoxia. Chest. 2012 Jun;141(6):1422-1430. doi: 10.1378/chest.11-1809. Epub 2012 Jan 5. PMID 22222188
- [Background] Perl J, Unruh ML, Chan CT. Sleep disorders in end-stage renal disease: 'Markers of inadequate dialysis'? Kidney Int. 2006 Nov;70(10):1687-93. doi: 10.1038/sj.ki.5001791. Epub 2006 Sep 13. PMID 16969388
- [Background] Hanly PJ, Ahmed SB. Sleep apnea and the kidney: is sleep apnea a risk factor for chronic kidney disease? Chest. 2014 Oct;146(4):1114-1122. doi: 10.1378/chest.14-0596. PMID 25288001
- [Background] Beecroft J, Duffin J, Pierratos A, Chan CT, McFarlane P, Hanly PJ. Enhanced chemo-responsiveness in patients with sleep apnoea and end-stage renal disease. Eur Respir J. 2006 Jul;28(1):151-8. doi: 10.1183/09031936.06.00075405. Epub 2006 Mar 1. PMID 16510459
- [Background] Faulx MD, Storfer-Isser A, Kirchner HL, Jenny NS, Tracy RP, Redline S. Obstructive sleep apnea is associated with increased urinary albumin excretion. Sleep. 2007 Jul;30(7):923-9. doi: 10.1093/sleep/30.7.923. PMID 17682664
- [Background] Zoccali C, Mallamaci F, Tripepi G. Nocturnal hypoxemia predicts incident cardiovascular complications in dialysis patients. J Am Soc Nephrol. 2002 Mar;13(3):729-733. doi: 10.1681/ASN.V133729. PMID 11856778
- [Background] Nicholl DD, Hanly PJ, Poulin MJ, Handley GB, Hemmelgarn BR, Sola DY, Ahmed SB. Evaluation of continuous positive airway pressure therapy on renin-angiotensin system activity in obstructive sleep apnea. Am J Respir Crit Care Med. 2014 Sep 1;190(5):572-80. doi: 10.1164/rccm.201403-0526OC. PMID 25033250
- [Background] Kuzniar TJ, Klinger M. Sleep apnea, continuous positive airway pressure, and renal health. Am J Respir Crit Care Med. 2014 Sep 1;190(5):486-7. doi: 10.1164/rccm.201407-1359ED. No abstract available. PMID 25171309
- [Background] Ahmed SB, Ronksley PE, Hemmelgarn BR, Tsai WH, Manns BJ, Tonelli M, Klarenbach SW, Chin R, Clement FM, Hanly PJ. Nocturnal hypoxia and loss of kidney function. PLoS One. 2011 Apr 29;6(4):e19029. doi: 10.1371/journal.pone.0019029. PMID 21559506
- [Background] Sakaguchi Y, Hatta T, Hayashi T, Shoji T, Suzuki A, Tomida K, Okada N, Rakugi H, Isaka Y, Tsubakihara Y. Association of nocturnal hypoxemia with progression of CKD. Clin J Am Soc Nephrol. 2013 Sep;8(9):1502-7. doi: 10.2215/CJN.11931112. Epub 2013 Jun 6. PMID 23744006
- [Background] Gottlieb DJ, Punjabi NM, Mehra R, Patel SR, Quan SF, Babineau DC, Tracy RP, Rueschman M, Blumenthal RS, Lewis EF, Bhatt DL, Redline S. CPAP versus oxygen in obstructive sleep apnea. N Engl J Med. 2014 Jun 12;370(24):2276-85. doi: 10.1056/NEJMoa1306766. PMID 24918372
- [Background] Mansfield DR, Gollogly NC, Kaye DM, Richardson M, Bergin P, Naughton MT. Controlled trial of continuous positive airway pressure in obstructive sleep apnea and heart failure. Am J Respir Crit Care Med. 2004 Feb 1;169(3):361-6. doi: 10.1164/rccm.200306-752OC. Epub 2003 Nov 3. PMID 14597482
- [Background] Koga S, Ikeda S, Yasunaga T, Nakata T, Maemura K. Effects of nasal continuous positive airway pressure on the glomerular filtration rate in patients with obstructive sleep apnea syndrome. Intern Med. 2013;52(3):345-9. doi: 10.2169/internalmedicine.52.8468. Epub 2013 Feb 1. PMID 23370742
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Levey AS, Inker LA, Matsushita K, Greene T, Willis K, Lewis E, de Zeeuw D, Cheung AK, Coresh J. GFR decline as an end point for clinical trials in CKD: a scientific workshop sponsored by the National Kidney Foundation and the US Food and Drug Administration. Am J Kidney Dis. 2014 Dec;64(6):821-35. doi: 10.1053/j.ajkd.2014.07.030. Epub 2014 Oct 16. PMID 25441437
- [Background] Inker LA, Lambers Heerspink HJ, Mondal H, Schmid CH, Tighiouart H, Noubary F, Coresh J, Greene T, Levey AS. GFR decline as an alternative end point to kidney failure in clinical trials: a meta-analysis of treatment effects from 37 randomized trials. Am J Kidney Dis. 2014 Dec;64(6):848-59. doi: 10.1053/j.ajkd.2014.08.017. Epub 2014 Oct 16. PMID 25441438
- [Background] Greene T, Teng CC, Inker LA, Redd A, Ying J, Woodward M, Coresh J, Levey AS. Utility and validity of estimated GFR-based surrogate time-to-event end points in CKD: a simulation study. Am J Kidney Dis. 2014 Dec;64(6):867-79. doi: 10.1053/j.ajkd.2014.08.019. Epub 2014 Oct 31. PMID 25441440
- [Background] Vigil A, Condes E, Vigil L, Gallar P, Oliet A, Ortega O, Rodriguez I, Ortiz M, Herrero JC, Mon C, Cobo G, Jimenez J. Cystatin C as a predictor of mortality and cardiovascular events in a population with chronic kidney disease. Int J Nephrol. 2014;2014:127943. doi: 10.1155/2014/127943. Epub 2014 Feb 11. PMID 24672725